CLINICAL TRIAL: NCT04585763
Title: Prospective, Multi-center, Single-arm Study of the Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL) System in Calcified Peripheral Arteries
Brief Title: Disrupt PAD+ Study With the Shockwave Medical M5+ Peripheral IVL System
Acronym: Disrupt PAD+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 64007
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Arterial Disease; Vascular Disease, Peripheral
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL) (Experimental)
  Interventions: Device: Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)

INTERVENTIONS:
Device: Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL) — The Shockwave Medical M5+ Peripheral IVL System is indicated for lithotripsy-enhanced, low-pressure balloon dilatation of lesions, including calcified lesions, in the peripheral vasculature, including the iliac, femoral, ilio-femoral, popliteal, infra-popliteal, and renal arteries. This device is not intended for use in coronary, carotid, or cerebrovascular arteries.

SUMMARY:
Prospective, multi-center, single-arm study of the M5+ Peripheral IVL system to treat calcified peripheral arteries.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety and performance of the Shockwave M5+ Peripheral IVL System to treat calcified peripheral arteries in pre-market countries, and to assess continued safety and effectiveness in the US. A minimum of 40 lesions in up to 40 subjects at up to 10 sites in Australia, New Zealand and the US will be enrolled with the aim of treating at least 20 target lesions with the 8.0 mm IVL catheter. A maximum of three target lesions may be treated per subject. Subjects with moderate and severely calcified iliac and femoropopliteal artery disease presenting with Rutherford Category 2 to 5. Approximately 6 months of enrollment at up to 10 sites in Australia, New Zealand and the US. Study subjects will be followed through discharge, 30 days, 6 and 12 months. Duplex Ultrasound (DUS) assessments will be completed at 12 months. Total anticipated study duration is 18 months. The primary safety endpoint is Major Adverse Events (MAE) at 30 days defined as: need for emergency surgical revascularization of target limb; unplanned target limb major amputation (above the ankle); symptomatic thrombus or distal emboli that require surgical, mechanical or pharmacologic means to improve flow and extend hospitalization ; or perforations that require an intervention, including bail-out stenting. The primary performance endpoint is technical success defined as final residual stenosis ≤30% without flow-limiting dissection (≥ Grade D) of the lesion by angiographic core lab.

ELIGIBILITY:
General Inclusion Criteria

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
3. Age of subject is > 18.
4. Rutherford Clinical Category 2, 3, 4 or 5 of the target limb(s).
5. Estimated life expectancy >1 year.
6. Subject is intended to undergo treatment with Shockwave M5+ Peripheral IVL System for de novo lesions of the ilio-femoropopliteal arteries.

   Angiographic Inclusion Criteria
7. Single or multiple de novo target lesion(s) located from the common iliac to the femoropopliteal artery, in one or both limbs.
8. Target lesion reference vessel diameter is between 3.5mm and 8.0mm by visual estimate.
9. Target lesion is ≥70% stenosis by investigator via visual estimate.
10. Target lesion length is ≤200mm for lesions 70-99% stenosed. Target lesion can be all or part of the 200mm treated zone.
11. Chronic total occlusion, lesion length is ≤100mm of the total ≤200 mm target lesion.
12. Subject has at least one patent tibial vessel on the target leg with runoff to the foot, defined as no stenosis >50%.
13. Calcification is at least moderate defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

General Exclusion Criteria

1. Rutherford Clinical Category 0, 1, and 6.
2. Subject has active infection requiring antibiotic therapy.
3. History of endovascular or surgical procedure on the target limb within the last 30 days or planned within 30 days of the index procedure. Note: Concomitant IVL treatment to facilitate large bore access at the time of procedure is allowed.
4. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
5. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
6. Subject has known allergy to urethane, nylon, or silicone.
7. Myocardial infarction within 60 days prior to enrollment.
8. History of stroke within 60 days prior to enrollment.
9. Subject has acute or chronic renal disease defined as serum creatinine of >2.5 mg/dL or >220 umol/L, unless on dialysis.
10. Subject is pregnant or nursing.
11. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
12. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
13. The planned use of specialty balloons, re-entry or atherectomy devices in the target lesion(s).

    Angiographic Exclusion Criteria
14. In-stent restenosis within 10mm of the target zone.
15. Target lesions distal to the popliteal artery.
16. Evidence of aneurysm or thrombus in target vessel.
17. No calcium or mild calcium in the target lesion.
18. Target lesion within native or synthetic vessel grafts.
19. Subject has more than three target lesions requiring treatment.
20. Subject has significant non-target lesion (>50% stenosis or occlusion) within the target limb (e.g. iliac, common femoral or below-the-knee) not successfully treated prior to treatment of the target lesions.
21. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - St. John Clinic, Bartlesville, Oklahoma
- Australia (2):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Perth Institute of Vascular Research, Nedlands, Western Australia
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato District Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Period: Overall Study
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Started | 37; 51 Lesions
Completed | 35; 48 Lesions
Not Completed | 2; 3 Lesions

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL): The Shockwave Medical M5+ Peripheral IVL System is indicated for lithotripsy-enhanced, low-pressure balloon dilatation of lesions, including calcified lesions, in the peripheral vasculature, including the iliac, femoral, ilio-femoral, popliteal, infra-popliteal, and renal arteries. This device is not intended for use in coronary, carotid, or cerebrovascular arteries.
Arm/Group | Single Arm
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 17
  United States | 10
  Australia | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: Defined as:
  Need for emergency surgical revascularization of target limb
  * Unplanned target limb major amputation (above the ankle)
  * Symptomatic thrombus or distal emboli that require surgical, mechanical or pharmacologic means to improve flow and extend hospitalization
  * Perforations that require an intervention, including bail-out stenting
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 37
Participants | 0

2. Primary Outcome: Number of Lesions With Technical Success
Description: Defined as final residual stenosis ≤30% without flow-limiting dissection (≥ Grade D) of the lesion by angiographic core lab.
Time Frame: Peri-procedural, approximately 2 hours
Population: Technical success is on a per lesion basis, not per subject.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 48
Number analyzed (Lesions) | 48
Lesions | 43

3. Secondary Outcome: Number of Lesions With IVL Technical Success
Description: Defined as residual stenosis ≤30% without flow-limiting dissection (≥ Grade D) of the lesion post-IVL by angiographic core lab
Time Frame: Peri-procedural, approximately 2 hours
Population: IVL Technical Success was calculated on a per lesion basis, not per subject.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 47
Number analyzed (Lesions) | 47
Lesions | 28

4. Secondary Outcome: Number of Participants With Procedural Success
Description: Defined as final residual stenosis ≤30% without any flow-limiting dissection (≥ Grade D) in all target lesions by angiographic core lab
Time Frame: Peri-procedural, approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 35
Participants | 30

5. Secondary Outcome: Number of Participants With Clinically-driven Target Lesion Revascularization (TLR)
Description: A target lesion revascularization performed due to target lesion diameter stenosis ≥50% and either evidence of clinical or functional ischemia (e.g., recurrent/progressive life-limiting intermittent claudication, claudication unresponsive to medical therapy, CLI) or recurrence of the clinical syndrome for which the initial procedure was performed. Clinically driven target lesion revascularization occurs in the absence of protocol directed surveillance ultrasound or angiography.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 37
Participants | 0

6. Secondary Outcome: Rutherford Category Reported as Change From Baseline
Description: Number of Participants with Improvement in Rutherford Score from as reported at 30 days post-procedure
Time Frame: 30 days
Population: Improved from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 32
Participants | 27

7. Secondary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: * Need for emergency surgical revascularization of target limb
  * Unplanned target limb major amputation (above the ankle)
  * Symptomatic thrombus or distal emboli that require surgical, mechanical or pharmacologic means to improve flow and extend hospitalization
  * Perforations that require an intervention, including bail-out stenting
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 37
Participants | 1

8. Secondary Outcome: Number of Participants With Clinically-driven Target Lesion Revascularization (TLR)
Description: as for outcome 5
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 37
Participants | 0

9. Secondary Outcome: Rutherford Category Reported as Change From Baseline
Description: Number of Participants with Improvement in Rutherford Score from as reported at 6 months post-procedure
Time Frame: 6 months
Population: Improved from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 34
Participants | 26

10. Secondary Outcome: Number of Participants With Primary Patency
Description: Defined as freedom from clinically-driven target lesion revascularization (TLR) and freedom from restenosis determined by duplex ultrasound or angiogram ≥50% stenosis
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 30
Participants | 21

11. Secondary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: as for outcome 7
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 35
Participants | 1

12. Secondary Outcome: Number of Participants With Clinically-driven Target Lesion Revascularization (TLR)
Description: as for outcome 5
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 35
Participants | 3

13. Secondary Outcome: Ankle-brachial Index (ABI) Reported as Change From Baseline
Description: ABI at 12 months reported as change from baseline. The ABI is the ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery. Ideally, this ratio should be 1.0, but is often less in a subject with peripheral arterial disease.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 24
ratio | 0.3 (0.5)

14. Secondary Outcome: Rutherford Category Reported as Change From Baseline
Description: Number of Participants with Improvement in Rutherford Score from as reported at 12 Months post-procedure.
Time Frame: 12 months
Population: Improved from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5+ Peripheral Intravascular Lithotripsy (IVL)
Number analyzed (Participants) | 32
Participants | 24

ADVERSE EVENTS:
Time Frame: This accounting is for all study events through the 12 month time frame.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 20/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=37)
Neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Pulmonary oedema (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastroinstestinal haemorrhage (Gastrointestinal disorders) | 1
Complication of device removal (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Biliary sepsis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Cholecystitis infective (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Nephropathy toxic (Injury, poisoning and procedural complications) | 1
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Leg amputation (Surgical and medical procedures) | 1
Rehabilitation therapy (Surgical and medical procedures) | 1
Arterial bypass stenosis (Vascular disorders) | 1
Blue toe syndrome (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Intermittent claudication (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 4
Peripheral artery dissection (Vascular disorders) | 4
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Retroperitoneal haemorrhage (Vascular disorders) | 1
Venous ulcer pain (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=37)
Atrial fibrillation (Cardiac disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
COVID-19 (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 3
Limb injury (Injury, poisoning and procedural complications) | 3
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Iliac artery dissection (Vascular disorders) | 2
Peripheral artery restenosis (Vascular disorders) | 6
Peripheral artery stenosis (Vascular disorders) | 3
Intermittent claudication (Vascular disorders) | 10
Peripheral arterial occlusive disease (Vascular disorders) | 4
Peripheral artery dissection (Vascular disorders) | 13
Ischemic rest pain (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT04585763/Prot_SAP_000.pdf